CLINICAL TRIAL: NCT01695382
Title: Apoyo Con Carino: Patient Navigation to Improve Palliative Care Outcomes for Latinos With Advanced Cancer
Brief Title: Apoyo Con Carino: Patient Navigation for Palliative Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 12-0592
Record Dates: First submitted 2012-09-25; First posted 2012-09-28 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Cancer
Keywords: Cancer; Palliative Care; Patient Navigation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Navigation (Experimental): Participants randomized to the control arm of the study will receive a packet of written materials that are appropriate linguistically and written for individuals with low health literacy. In addition they will have 5 navigator initiated home visits to review the educational materials and help patients and families address barriers to palliative care through education, advocacy, and activation.
  Interventions: Behavioral: Navigation
- Control (No Intervention): Participants randomized to the control arm of the study will receive a packet of written materials that are appropriate linguistically and written for individuals with low health literacy.

INTERVENTIONS:
Behavioral: Navigation — As per Arm description
  Arms: Navigation

SUMMARY:
Palliative care is a priority area of focus for health care in an aging population experiencing burdens of chronic illness. Despite the evidence-based benefits of palliative care, access remains limited, especially in poor urban and rural settings. Cultural and linguistic barriers may also increase disparities in palliative care for Latinos. Due to a nationwide shortage of palliative care providers and the unique cultural preferences and values of patients, the investigators are testing a patient navigator intervention to improve palliative care outcomes for Latinos with advanced cancer.

DETAILED DESCRIPTION:
This project uses a patient navigator to deliver a culturally tailored intervention to improve palliative care for Latinos with advanced cancer in urban and rural communities. The proposed research aims to improve palliative care with the goal of preventing and relieving suffering for people facing serious, complex illness. Palliative care, according to the National Quality Forum and Centers for Medicare and Medicaid, provides patient and family-centered care offered in conjunction with curative and all other appropriate forms of medical treatment. It addresses physical, intellectual, emotional, social, spiritual needs, and facilitates patients' understanding of illness and choice. There is emerging evidence that palliative care may also improve survival for cancer patients. The proposed research also focuses on reducing health disparities. Studies have shown that Latinos are more likely to die in a hospital, less likely to use hospice services, and more likely to have unmanaged pain. This study will recruit 240 Latino patients with advanced cancer from an urban safety net hospital, a National Cancer Institute-designated Comprehensive Cancer Center, and several rural communities (including some of the poorest, most underserved counties in Colorado). Patients will be randomized to either a control or intervention group. The control group will receive written materials covering three important palliative care domains -advance care planning, pain management, and hospice care. The materials, in English and Spanish, are appropriate for patients with low health literacy. Patients in the intervention group will receive the same written materials but will also have a patient navigator who will make 5 home visits to review materials, help patients and families talk about goals/values, and complete an advance directive, all in a culturally and linguistically appropriate manner. The navigator may also help with: accessing community resources, participating in family meetings with health care providers, and offering support to patients and families. The investigators hypothesize that the intervention will increase advance care planning, improve pain management, increase hospice referrals, and patients will have improved palliative care overall at the end of life. The patient navigator model has demonstrated an ability to improve cancer screening, early diagnosis, treatment, and survivorship. Once the investigators demonstrate the efficacy of a patient navigator intervention to improve palliative care for advanced cancer patients, they can disseminate the training and intervention to all patient navigators working with Latino cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Stage III or Stage IV cancer (all types)
* Self-identify as Latino
* 18 years of age or older
* Speak English or Spanish

Exclusion Criteria:

* Lacking decisional capacity
* Incarcerated

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Improvement in Palliative Care Overall | 3 months after enrollment
  Patient Navigator and Process Measure will capture the less tangible benefits of a patient navigator and help understand the effects of the many activities of the navigator beyond the scope of the prescribed intervention. The questions incorporate aspects of self-efficacy and patient activation (key concepts that patient navigators help improve).
Evidence of Advance Care Planning | 6 months after enrollment
  Chart review to determine if there is an advance directive in the medical record and classification of the type of advance directive (Medical Durable Power of Attorney (MDPOA), Advance Directive (AD), Living Will)
Assesment of Pain Management | 3 months after enrollment
  Pain management will be assessed through patient interviews utilizing the Brief Pain Inventory (BPI). The BPI Long Form (BPI-LF) is a 32-item self-report instrument that assesses the severity and impact of pain in patients with chronic diseases, e.g. cancer.
Hospice Utilization | 46 months after enrollment
  Length of stay in hospice program in days. Data will be collected through follow up phone calls, medical records review, and death records review to determine date of admission into hospice program and date of discharge (through death or dis-enrollment)

SECONDARY OUTCOMES:
Aggressiveness of Care at the End of Life | At month 46
  For patients who have died within the follow up period this outcome assesses aggressiveness of care at the end of life using a composite measure comprised of the following: chemotherapy within 14 days of death no hospice hospice within 3 days of death
Change in Quality of Life | Baseline and 3 months after enrollment
  McGill Quality of Life questionnaire (MQOL) will be used at baseline and at 3 months after enrollment. The MQOL is specifically designed for a palliative care population, measuring whole-person concerns magnified by advanced life-limiting illness. It is short, reliable, repeatable, and can be used to determine changes in QOL of groups.

CONTACTS AND LOCATIONS:
Overall Officials: Stacy M Fischer, MD, Principal Investigator — University of Colorado, Denver
Locations (5):
- United States (5):
  - San Luis Valley Regional Medical Center, Alamosa, Colorado
  - University of Colorado Cancer Center, Aurora, Colorado
  - Denver Health and Hospital Authority, Denver, Colorado
  - Shaw Cancer Center, Eagle, Colorado
  - Valley View Medical Center, Glenwood Springs, Colorado

REFERENCES:
- [Derived] Fischer SM, Kline DM, Min SJ, Okuyama-Sasaki S, Fink RM. Effect of Apoyo con Carino (Support With Caring) Trial of a Patient Navigator Intervention to Improve Palliative Care Outcomes for Latino Adults With Advanced Cancer: A Randomized Clinical Trial. JAMA Oncol. 2018 Dec 1;4(12):1736-1741. doi: 10.1001/jamaoncol.2018.4014. PMID 30326035
- [Derived] Fischer SM, Kline DM, Min SJ, Okuyama S, Fink RM. Apoyo con Carino: Strategies to Promote Recruiting, Enrolling, and Retaining Latinos in a Cancer Clinical Trial. J Natl Compr Canc Netw. 2017 Nov;15(11):1392-1399. doi: 10.6004/jnccn.2017.7005. PMID 29118231